CLINICAL TRIAL: NCT06314789
Title: The Role and Importance of Lung Ultrasound Score Used in the Delivery Room in the Early Diagnosis of Respiratory Morbidities in Newborns
Brief Title: The Use of Lung Ultrasonography in the Delivery Room in Neonates
Acronym: LUSIN
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Umran Koral, MD, Kırıkkale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: G1201
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Suspected Damage to Fetus From Other Disease in the Mother, Affecting Management of Mother, With Delivery; Patient Death or Serious Disability Associated With A Haemolytic Reaction Due to the Administration of ABO-Incompatible Blood or Blood Products
Keywords: newborn, premature infant, lung ultrasonography
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung ultrasound for newborns (Experimental): In the study, both LUS imaging and scoring will be performed in the delivery room within the first 30 minutes and lUS score evaluation will be performed at postnatal 2nd, 6th and 24th hours in the intensive care unit for inpatients and in the maternal ward for maternal patients.
  Interventions: Diagnostic Test: doing lung ultrasonography

INTERVENTIONS:
Diagnostic Test: doing lung ultrasonography — In the study, both LUS imaging and scoring will be performed in the delivery room within the first 30 minutes and LUS score evaluation will be performed at postnatal 2nd, 6th and 24th hours in the intensive care unit for inpatients and in the maternal ward for maternal patients.

SUMMARY:
Lung ultrasonography has become frequently used in neonatal intensive care units because it is a diagnostic, useful, harmless, radiation-free, bedside, reproducible and practical method. (1, 2) In our clinic, lung ultrasonography imaging is performed in infants hospitalized with respiratory distress.

Lung ultrasonography is widely used especially in conditions that mainly cause respiratory distress such as respiratory distress syndrome (RDS), pneumonia, neonatal transient tachypnea (NTRT), congenital pneumonia, meconium aspiration syndrome and pneumothorax. (1, 2) The reliability and specificity of AUS imaging especially in the diagnosis of NTRT have been proven in many studies.

AUS imaging has become an objective value by scoring today. Images will be obtained using the linear probe of the device to be used for lung ultrasound and transferred to a cell phone, both lungs will be evaluated as three areas on the right and left (anterior upper, anterior lower and lateral) and scored separately. Anteriorly, the region between the anterior axillary line and the parasternal line is divided into two by the line passing through the nipple. Above is considered as the upper anterior region and below as the lower anterior region. The area in the middle of the anterior and posterior axillary line is evaluated as the lateral region. Each area is scored from 0 to 3 points. If A lines are present, 0 points are given, if there are more than 3 B lines in an area, 1 point is given, if B lines are very dense and there are no A lines, it is considered as white lung and 2 points are given. If there is a consolidation image on AUS, 3 points were given. The maximum total score was 18 (8,9) (Figure 1).

In this study, both AUS imaging and scoring will be performed in the delivery room within the first 30 minutes and AUS score evaluation will be performed at postnatal 2nd, 6th and 24th hours in the intensive care unit for inpatients and in the maternal ward for maternal patients. The hypothesis of this study is that newborns with high AUS scores will have high rates of respiratory morbidities and respiratory support in the neonatal unit. The primary aim of the study was to determine the role and importance of AUS scores measured in the delivery room in predicting respiratory morbidities of infants. The secondary aim was to investigate the value of the course of AUS scores at postnatal 2, 6 and 24 hours in predicting the respiratory prognosis of the newborn infant.

DETAILED DESCRIPTION:
Lung ultrasonography (LUS) was first used in adults in 1995 and has been used in neonatology and pediatrics in recent years and has become increasingly widespread. Lung ultrasonography has become frequently used in neonatal intensive care units because it is a diagnostic, useful, harmless, radiation-free, bedside, reproducible and practical method. (1, 2) In our clinic, lung ultrasonography imaging is performed in infants hospitalized with respiratory distress.

Lung ultrasonography is widely used especially in conditions that mainly cause respiratory distress such as respiratory distress syndrome (RDS), pneumonia, neonatal transient tachypnea (NTRT), congenital pneumonia, meconium aspiration syndrome and pneumothorax. (1, 2) The reliability and specificity of AUS imaging especially in the diagnosis of RDS have been proven in many studies. (1,2,3) The diagnosis of RDS on lung ultrasonography is made by "visualization of the transition zone (double lung point)" (3). In addition, "white lung appearance" in RDS, "absence of pleural motion and "barcode" appearance in M mode" in the presence of pneumothorax, one of the air leakage syndromes, and "hepatization/consolidation appearance" in pneumonia are among ultrasonographic findings (1,3).

In infants whose lung ultrasound findings are compatible with RDS and who clinically require surfactant, surfactant therapy is given in a shorter time without waiting for chest radiography. In a study involving 40 patients diagnosed with RDS, it was found that there was a significant improvement ultrasonographically in the 4th hour of surfactant treatment, and in another study, it was shown that chest radiography was dramatically reduced with the use of AUS. (4, 5) In the light of this information, we see that the use of AUS is becoming increasingly widespread in newborns. AUS imaging has now become an objective value by scoring. With these scores, the relationship between the diagnosis of the disease and the score has been tried to be determined and related studies have been conducted. (6,7) Images will be obtained using the linear probe of the device to be used for lung ultrasound and transferred to a cell phone. The AUS scoring described in the studies of Brat et al. and Raimondi et al. (8,9) Accordingly, both lungs will be evaluated as three areas on the right and left (anterior superior, anterior inferior and lateral) and scored separately. Anteriorly, the region between the anterior axillary line and the parasternal line is divided into two by the line passing through the nipple. Above is considered as the upper anterior region and below as the lower anterior region. The area in the middle of the anterior and posterior axillary line is evaluated as the lateral region. Each area is scored from 0 to 3 points. If A lines are present, 0 points are given, if there are more than 3 B lines in an area, 1 point is given, if B lines are very dense and there are no A lines, it is considered as white lung and 2 points are given. If there is a consolidation image on AUS, 3 points were given. The maximum total score was 18 (8,9) (Figure 1).

The transition from fetal to extrauterine life requires numerous rapid organ adaptations. Clearance of fetal lung fluid, surfactant secretion and the onset of steady breathing occur during pulmonary adaptation, and changes in blood flow, increased cardiac output and pulmonary vasodilation occur for the cardiovascular transition. (10) This period typically lasts for two hours. During this period, placental breathing is replaced by spontaneous breathing. When there is a delay in transition during this adaptation process, tachypnea and moaning may be observed. This process should be distinguished from transient tachypnea (wet lung) of the newborn. In case of respiratory distress that persists after the first two hours postnatally, the transition delay is avoided (10). Transient tachypnea of the newborn is considered as a possible diagnosis. If there is a risk factor or respiratory distress persists and laboratory and imaging methods support it, congenital pneumonia at 34 weeks and above is frequently included among the diagnoses presenting with respiratory distress. In addition, RDS can also be seen rarely in this period (3).

When we perform AUS imaging in the delivery room, i.e. within the first 30 minutes, we may see pulmonary edema, diffuse B lines, or a normal lung that has completed its transition and has more A lines. Newborns who do not require neonatal hospitalization due to respiratory distress will also be followed up in the maternal ward and their clinic will be evaluated according to the AUS score they received in the delivery room.

In the study, both AUS imaging and scoring will be performed in the delivery room within the first 30 minutes and AUS score evaluation will be performed in the intensive care unit for inpatients and in the maternity ward for maternal patients at postnatal 2nd, 6th and 24th hours. The hypothesis of this study is that newborns with high AUS scores will have high rates of respiratory morbidities and respiratory support in the neonatal unit. The primary aim of the study was to determine the role and importance of AUS scores measured in the delivery room in predicting respiratory morbidities of infants. The secondary aim was to investigate the value of the course of AUS scores at postnatal 2, 6 and 24 hours in predicting the respiratory prognosis of the newborn infant.

Sources:

1. Raimondi F, Cattarossi L, Copetti R. Point-of-care chest ultrasound in the neonatal intensive care unit: an Italian Perspective. Neoreviews 2014;15:e2-6.
2. Escourrou G., De Luca D. Lung ultrasound decreased radiation exposure in preterm infants in a neonatal intensive care unit. Acta Pediatrica 2016; e237-e239.
3. Raimondi F. et al. A Multicenter Lung Ultrasound Study on Transient Tachypnea of the Neonate. Neonatology 2019; 115:263-268
4. Oktem A, Yigit S, Oğuz B, Celik T, Haliloğlu M, Yurdakok M. Accuracy of Lung Ultrasonography in the Diagnosis of Respiratory Distress Syndrome in Newborns. J Matern Fetal Neonatal Med. 2019 Apr 22;1-6.
5. Tandircioglu UA, Yigit S, Oguz B, Kayki G, Celik HT, Yurdakok M. Lung ultrasonography decreases radiation exposure in newborns with respiratory distress: a retrospective cohort study. Eur J Pediatr. 2022 Mar;181(3):1029-1035. doi: 10.1007/s00431-021-04296-5.
6. Liu J. The Lung Ultrasound Score Cannot Accurately Evaluate the Severity of Neonatal Lung Disease. J Ultrasound Med. 2020 May;39(5):1015-1020. doi: 10.1002/jum.15176. Epub 2019 Nov 18. PMID: 31737918.
7. Pang H, Zhang B, Shi J, Zang J, Qiu L. Diagnostic value of lung ultrasound in evaluating the severity of neonatal respiratory distress syndrome. Eur J Radiol. 2019 Jul;116:186-191. doi: 10.1016/j.ejrad.2019.05.004.
8. Brat R, Yousef N, Klifa R, Reynaud S, Shankar Aguilera S, De Luca D. Lung ultrasonography score to evaluate oxygenation and surfactant need in neonates treated with continuous positive airway pressure. JAMA Pediatr. 2015;169(8):e151797
9. Raimondi F, Migliaro F, Corsini I, et al. Lung Ultrasound Score Progress in Neonatal Respiratory Distress Syndrome. Pediatrics. 2021;147(4):e2020030528
10. Hillman NH, Kallapur SG, Jobe AH. Physiology of transition from intrauterine to extrauterine life. Clin Perinatol. 2012;39(4):769-83.
11. Poerio A, Galletti S, Baldazzi M, Martini S, Rollo A, Spinedi S, et al. Lung ultrasound features predict admission to the neonatal intensive care unit in infants with transient neonatal tachypnoea or respiratory distress syndrome born by caesarean section. Eur J Pediatr. 2021 Mar;180(3):869-876. doi: 10.1007/s00431-020-03789-z.

ELIGIBILITY:
Inclusion Criteria:

* Patients born in Kırıkkale University Faculty of Medicine Hospital who were over 34 weeks and who underwent lung ultrasonography from the delivery room
* Patients who consented to the study

Exclusion Criteria:

* Patients born under 34 weeks
* Patients whose delivery did not take place at Kırıkkale University Medical Faculty Hospital
* Patients without study consent
* Patients with lung anomalies
* Congenital heart disease
* Those with major congenital anomalies

Ages: 1 Minute to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 112 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
LUS in delivery room | 0-30 minutes
  Predicting respiratory morbidities in newborns with lung ultrasound score performed in the delivery room

SECONDARY OUTCOMES:
LUS in NICU or room | 24 hours
  Predicting the severity of respiratory morbidities with repeated AUS scores.

CONTACTS AND LOCATIONS:
Overall Officials: Umit Ayse Tandircioglu, Principal Investigator — Kırıkkale University
Locations (1):
- Kirikkale University, Kırıkkale, Turkey (Türkiye)